CLINICAL TRIAL: NCT05928065
Title: Ultrasound Analysis of Suspected Long Bone Fractures in the Emergency Department - Diagnostic Performance Compared to Radiography.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1422021/CHUSTE
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Bone Fracture
Keywords: bone trauma; bone; Ultrasound; fracture; radiography
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with low kinetic, non-deforming, non-open long bone trauma: Children with low kinetic, non-deforming, non-open long bone trauma will be included.
  Collection of datas of medical record.
  Interventions: Other: Collection of datas

INTERVENTIONS:
Other: Collection of datas — Collection of datas: datas of physical examination (swelling, hematoma, edema), benign trauma (non deforming and closed fractures), ultrasound and radiographic images and evaluation of pain.

SUMMARY:
Ultrasound tool in bones trauma is underused in the emergency department of the University Hospital of Saint-Etienne. This prospective non randomized monocentric study will measure how much this non irradiant method of diagnostic is sensible and specific in long bones fractures, and will evaluate it advantages versus conventional X ray examination.

DETAILED DESCRIPTION:
This study is based on physical examination (swelling, hematoma, edema) and concerns all long bones, including benign trauma (non deforming and closed fractures). The necessary time to make an ultrasound conclusion and the operator certitude degree will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Children with low kinetic, non-deforming, non-open long bone trauma

Exclusion Criteria:

* Opened fracture, deforming trauma

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged between 0 to 18 with low kinetic, non-deforming, non-open long bone trauma will be included.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Analysis concordance between the ultrasound and radiographic method for the diagnosis of long bone fractures. | Year: 1
  Analysis datas collected.

SECONDARY OUTCOMES:
Analysis diagnostic performance between the ultrasound and radiographic method | Year: 1
  Analysis datas collected.

CONTACTS AND LOCATIONS:
Overall Officials: Aymeric CANTAIS, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No